CLINICAL TRIAL: NCT02213861
Title: A Randomized Phase 2 Study to Evaluate Three Treatment Regimens of SHAPE, a Histone Deacetylase Inhibitor, in Patients With Stage IA, IB or IIA Cutaneous T-Cell Lymphoma
Brief Title: Efficacy, Safety and Tolerability Study of SHAPE in IA, IB or IIA Cutaneous T-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: TetraLogic Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHP-141-003
Record Dates: First submitted 2014-08-06; First posted 2014-08-12 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Cutaneous T-Cell Lymphoma (CTCL)
Keywords: CTCL; Cutaneous T-Cell Lymphoma; Early-stage; SHAPE; SHP-141; topical; Histone deacetylase inhibitor; CAILS; mSWAT; mycosis fungoides
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1.0% SHAPE Gelled Solution once daily (Experimental)
  Interventions: Drug: SHAPE
- 0.5% SHAPE Gelled Solution twice daily (Experimental)
  Interventions: Drug: SHAPE
- 1.0% SHAPE Gelled Solution twice daily (Experimental)
  Interventions: Drug: SHAPE

INTERVENTIONS:
Drug: SHAPE — topical gel
  Other Names: SHP-141

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of SHAPE administered topically to skin lesions in patients with early-stage cutaneous T-cell lymphoma (CTCL).

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, open-label, randomized study to evaluate the efficacy and safety of SHAPE Gelled Solution applied topically daily or twice daily for 26 consecutive weeks to specified skin lesions in patients with Stage IA, IB or IIA CTCL. Patients responding to treatment will be allowed to continue on study for a maximum of 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of CTCL; a documented verifiable biopsy report is required
* Documented clinical stage IA, IB or IIA CTCL
* Skin lesion involvement of at least 2% of BSA accessible for topical application of study drug
* ECOG performance status of 0-2

Exclusion Criteria:

* CTCL with histologic evidence of folliculotropic variant or large cell transformed CTCL
* Palpable lymph node ≥1.5 cm in diameter (unless the lymph node has been biopsied and designated as Stage IA-IIA disease)
* Co-existent second malignancy or history of prior solid organ malignancy within previous 5 years (excluding basal or squamous cell carcinoma, in situ carcinoma of the cervix (CIN3), papillary or follicular thyroid cancer or prostate cancer that has been treated curatively
* Any prior history of hematologic malignancy (other than CTCL) within past 5 years
* CTCL disease that is known to be refractory to systemic histone deacetylase inhibitors
* Prior or concurrent central nervous system (CNS) metastases
* History of or current major gastrointestinal, pulmonary, cardiovascular, genitourinary or hematologic disease, CNS disorders, infectious disease or coagulation disorders as determined by the Investigator
* Evidence of active Hepatitis B or C or HIV
* Circulating atypical cells of clinical significance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Lesion severity using CAILS (Composite Assessment of Index Lesion Severity) | Every 4 weeks for 26 weeks and every 4 weeks thereafter for patients who continue on study (up to 52 weeks).

SECONDARY OUTCOMES:
modified Severity Weighted Assessment Tool (mSWAT) | Every 4 weeks for 26 weeks and every 4 weeks therafter for patients who continue on study (up to 52 weeks).
Patient assessment of pruritis using a Visual Analog Scale (VAS) | Every 4 weeks for 26 weeks and every 4 weeks thereafter for patients who continue on study (up to 52 weeks).
Skindex-29 Quality of Life Tool | Every 4 weeks for 26 weeks
modified Composite Assessment of Index Lesion Severity (CAILS) | Every 4 weeks for 26 weeks and every 4 weeks therafter for patients who continue on study (up to 52 weeks).

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Stanford Cancer Center, Stanford, California
  - Northwestern Medical Group, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Valipour A, Jager M, Wu P, Schmitt J, Bunch C, Weberschock T. Interventions for mycosis fungoides. Cochrane Database Syst Rev. 2020 Jul 7;7(7):CD008946. doi: 10.1002/14651858.CD008946.pub3. PMID 32632956